CLINICAL TRIAL: NCT04484337
Title: A Phase 1, Two-part, Double-blind, Active-control, Randomized Study to Evaluate the Pharmacokinetics, Safety and Tolerability of Repeat-Dose Cabotegravir (CAB 400 mg/mL Formulation) Long-Acting Injection Following Subcutaneous or Intramuscular Administration in Healthy Adult Participants
Brief Title: Study to Evaluate Pharmacokinetic (PK), Safety and Tolerability of Cabotegravir (CAB) 400 Milligrams Per Milliliter (mg/mL) Formulation in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 212482
Record Dates: First submitted 2020-07-20; First posted 2020-07-23 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: HIV Infections
Keywords: Cabotegravir; Long-Acting Injection; Pharmacokinetics; Safety; Tolerability
MeSH Terms: conditions — HIV Infections | interventions — cabotegravir; Lead; Anti-Inflammatory Agents, Non-Steroidal; Steroids

STUDY DESIGN:
Intervention Model Description: Participants will receive repeat doses of long-acting CAB 400 mg/mL or CAB 200 mg/mL at four-weekly (Q4W) interval in Part 1 and at 12-weekly (Q12W) interval in Part 2.
Who Masked: Participant, Investigator
Masking Description: This will be a double-blind (sponsor-unblind) study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (15):
- Part 1:Cohort 1: CAB 400 mg/mL IM gluteal (Experimental)
  Interventions: Drug: Cabotegravir sodium (Oral Lead In); Drug: Cabotegravir 400 mg/mL
- Part 1:Cohort 1: CAB 200 mg/mL IM gluteal (Active Comparator)
  Interventions: Drug: Cabotegravir sodium (Oral Lead In); Drug: Cabotegravir 200 mg/mL
- Part 1:Cohort 2: CAB 400 mg/mL SC abdominal (Experimental)
  Interventions: Drug: Cabotegravir sodium (Oral Lead In); Drug: Cabotegravir 400 mg/mL
- Part 1:Cohort 2: CAB 200 mg/mL SC abdominal (Active Comparator)
  Interventions: Drug: Cabotegravir sodium (Oral Lead In); Drug: Cabotegravir 200 mg/mL
- Part 1:Cohort 3: CAB 400 mg/mL IM (lateral thigh) (Experimental)
  Interventions: Drug: Cabotegravir sodium (Oral Lead In); Drug: Cabotegravir 400 mg/mL
- Part 1:Cohort 3: CAB 200 mg/mL IM (lateral thigh) (Active Comparator)
  Interventions: Drug: Cabotegravir sodium (Oral Lead In); Drug: Cabotegravir 200 mg/mL
- Part 1: Cohort 4: CAB 400 mg/mL (IM or SC) (Experimental)
  Interventions: Drug: Cabotegravir sodium (Oral Lead In); Drug: Cabotegravir 400 mg/mL
- Part 1: Cohort 4: CAB 200 mg/mL (IM or SC) (Active Comparator)
  Interventions: Drug: Cabotegravir sodium (Oral Lead In); Drug: Cabotegravir 200 mg/mL
- Part 2: Cohort 5: CAB 400 mg/mL IM (gluteus medius) (Experimental)
  Interventions: Drug: Cabotegravir sodium (Oral Lead In); Drug: Cabotegravir 400 mg/mL
- Part 2: Cohort 5: CAB 200 mg/mL IM (gluteus medius) (Active Comparator)
  Interventions: Drug: Cabotegravir sodium (Oral Lead In); Drug: Cabotegravir 200 mg/mL
- Part 2: Cohort 6: CAB 400 mg/mL IM (gluteus medius) (Experimental)
  Interventions: Drug: Cabotegravir sodium (Oral Lead In); Drug: Cabotegravir 400 mg/mL
- Part 2: Cohort 6: CAB 200 mg/mL IM (gluteus medius) (Active Comparator)
  Interventions: Drug: Cabotegravir sodium (Oral Lead In); Drug: Cabotegravir 200 mg/mL
- Part 1: Cohort 4b: CAB 400 mg/mL (SC) (Experimental)
  Interventions: Drug: Cabotegravir sodium (Oral Lead In); Drug: Cabotegravir 400 mg/mL; Drug: Topical non-steroidal anti-inflammatory drug; Drug: Topical steroid; Drug: Placebo creams/gels
- Part 1: Cohort 4h: CAB 400 mg/mL (SC) (Experimental)
  Interventions: Drug: Cabotegravir sodium (Oral Lead In); Drug: Cabotegravir 400 mg/mL; Drug: Recombinant human hyaluronidase PH20 (rHuPH20)
- Part 1: Cohort 4h: CAB 200 mg/mL (SC) (Active Comparator)
  Interventions: Drug: Cabotegravir sodium (Oral Lead In); Drug: Cabotegravir 200 mg/mL; Drug: Recombinant human hyaluronidase PH20 (rHuPH20)

INTERVENTIONS:
Drug: Cabotegravir sodium (Oral Lead In) — CAB will be available as 30 mg tablets for oral administration.
Drug: Cabotegravir 400 mg/mL — CAB 400 mg/mL will be available for administration by IM injection or SC Injection.
  Arms: Part 1: Cohort 4: CAB 400 mg/mL (IM or SC); Part 1: Cohort 4b: CAB 400 mg/mL (SC); Part 1: Cohort 4h: CAB 400 mg/mL (SC); Part 1:Cohort 1: CAB 400 mg/mL IM gluteal; Part 1:Cohort 2: CAB 400 mg/mL SC abdominal; Part 1:Cohort 3: CAB 400 mg/mL IM (lateral thigh); Part 2: Cohort 5: CAB 400 mg/mL IM (gluteus medius); Part 2: Cohort 6: CAB 400 mg/mL IM (gluteus medius)
Drug: Cabotegravir 200 mg/mL — CAB 200 mg/mL will be available for administration by IM injection or SC Injection.
  Arms: Part 1: Cohort 4: CAB 200 mg/mL (IM or SC); Part 1: Cohort 4h: CAB 200 mg/mL (SC); Part 1:Cohort 1: CAB 200 mg/mL IM gluteal; Part 1:Cohort 2: CAB 200 mg/mL SC abdominal; Part 1:Cohort 3: CAB 200 mg/mL IM (lateral thigh); Part 2: Cohort 5: CAB 200 mg/mL IM (gluteus medius); Part 2: Cohort 6: CAB 200 mg/mL IM (gluteus medius)
Drug: Topical non-steroidal anti-inflammatory drug — Non-steroidal anti-inflammatory drug will be available for topical application
  Arms: Part 1: Cohort 4b: CAB 400 mg/mL (SC)
Drug: Topical steroid — Steroid will be available for topical application
  Arms: Part 1: Cohort 4b: CAB 400 mg/mL (SC)
Drug: Placebo creams/gels — Placebo creams/gels will be available for topical application
  Arms: Part 1: Cohort 4b: CAB 400 mg/mL (SC)
Drug: Recombinant human hyaluronidase PH20 (rHuPH20) — rHuPH20 will be available for administration by SC Injection
  Arms: Part 1: Cohort 4h: CAB 200 mg/mL (SC); Part 1: Cohort 4h: CAB 400 mg/mL (SC)

SUMMARY:
This is an active control, randomized study to investigate the safety, tolerability and PK of repeat dose administration of long-acting CAB 400 mg/mL formulation intramuscular (IM) (gluteus medius and vastus lateralis) and subcutaneous (SC) (abdominal) injections in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 50 years of age inclusive, at the time of signing the informed consent.
* Participants who are overtly healthy as determined by medical evaluation.
* A participant with a clinical abnormality or laboratory parameters which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included if the investigator determines and documents that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Participants who are negative on two consecutive tests for Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), performed at Screening and within 5 days of admission to the Phase I unit, using an approved molecular test (Polymerase chain reaction [PCR]).
* Body weight more than or equal to (>=)40 kilogram (kg) and body mass index (BMI) within the range 18 to 32 kilogram per square meter (kg/m^2).
* Male participants are eligible to participate if they agree to use contraceptive methods and refrain from donating sperm.
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies: Is not a woman of childbearing potential (WOCBP) or is a WOCBP and using a contraceptive method that is highly effective, with a failure rate of less than (<)1 percent(%).
* Capable of giving signed informed consent.

Exclusion Criteria:

* Signs and symptoms which in the opinion of the investigator are suggestive of Coronavirus disease 2019 (COVID-19) (that is [i.e.] fever, cough etc) within 14 days of inpatient admission.
* Contact with known COVID-19 positive person/s in the 14 days prior to inpatient admission.
* History or presence of/significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention or interfering with the interpretation of data.
* Abnormal blood pressure as determined by the investigator.
* Alanine transaminase (ALT) more than (>)1.5 times upper limit of normal (ULN).
* Bilirubin >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Corrected QT interval (QTc) >450 milliseconds (msec).
* A known hypersensitivity to hyaluronidases (Cohort 4h only).
* The participant has an underlying skin disease or disorder (infection, inflammation, dermatitis, eczema, drug rash, drug allergy, psoriasis, food allergy, urticaria) that would interfere with assessment of injection sites.
* Current or anticipated need for chronic anti-coagulation with the exception of the use of low dose acetylsalicylic acid (less than or equal to [<=]325 mg) or hereditary coagulation and platelet disorders such as hemophilia or Von Willebrand Disease.
* Participants considered to have insufficient musculature to allow safe administration of CAB 400 mg/mL (gluteus medius or vastus lateralis).
* History of ongoing or clinically relevant seizure disorder within the previous 2 years, including participants who have required treatment for seizures within this time period.
* History of or on-going high-risk behaviors that may put the participant at increased risk for Human Immunodeficiency Virus (HIV) acquisition in the opinion of the investigator. This includes participants in HIV discordant relationships, or men who report current or prior unprotected anal sex with other men and those reporting prior or current injecting drug use.
* Participation in another concurrent clinical study or prior clinical study (with the exception of imaging trials) prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Participation in the study would result in loss of blood or blood products in excess of 500 mL within 56 days.
* The participant has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Presence of hepatitis B surface antigen (HBsAg), or positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment.
* A positive pre-study drug/alcohol screen.
* Exclusion criteria for screening electrocardiogram (ECG):

  1. Heart rate: For Males <45 or >100 beats per minute (bpm), for females <50 or >100 bpm.
  2. PR Interval: For males and females <120 or >220 msec.
  3. QRS duration: For males and females <70 or >120 msec.
  4. QT duration corrected for heart rate by Fridericia's formula (QTcF) interval: For males and females >450 msec.
* Evidence of previous myocardial infarction.
* Any conduction abnormality (including but not specific to left or right complete bundle branch block, atrioventricular [AV] block [2nd degree or higher], Wolff-Parkinson-White [WPW] syndrome).
* Sinus Pauses >3 seconds.
* Any significant arrhythmia which, in the opinion of the Investigator or GlaxoSmithKline (GSK)/ViiV Medical monitor, will interfere with the safety for the individual participant.
* Non-sustained or sustained ventricular tachycardia (>=3 consecutive ventricular ectopic beats).
* Positive HIV antibody/antigen test. Participants will be advised regarding safer sex. In the event a participant acquires HIV during the course of the study they will be required to withdraw from the study and will be referred urgently to an HIV treatment center for further management.
* Regular use of known drugs of abuse.
* Regular use of tobacco- or nicotine-containing products within 3 months prior to screening.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy.
* Participants with a history of intolerance to or with contraindications to the use of topical non-steroidal anti-inflammatory drugs (NSAIDs) or topical steroids will be excluded from participation in Cohort 4b.
* Regular alcohol consumption within 6 months prior to the study defined as: An average weekly intake of >14 units for males or >7 units for females.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products (e.g. nicotine patches or vaporizing devices) within 6 months prior to screening.
* The participant has a tattoo or other dermatological condition overlying the location of injection or a prior history of silicone implants (gluteal) which may interfere with interpretation of injection site reactions or administration of CAB LA.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 138 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
Maximum observed Plasma concentration (Cmax) for cabotegravir (Part 1 Injection 1) | Injection 1 Day 1 to Injection 1 Week 4
Cmax for cabotegravir (Part 1 Injection 2) | Injection 2 Day 1 to Week 52 follow-up
Cmax for cabotegravir (Part 2 Injection 1) | Injection 1 Day 1 to Injection 1 Week 12
Cmax for cabotegravir (Part 2 Injection 2) | Injection 2 Day 1 to Week 52 follow-up
Time of maximum observed plasma concentration (Tmax) for cabotegravir (Part 1 Injection 1) | Injection 1 Day 1 to Injection 1 Week 4
Tmax for cabotegravir (Part 1 Injection 2) | Injection 2 Day 1 to Week 52 follow-up
Tmax for cabotegravir (Part 2 Injection 1) | Injection 1 Day 1 to Injection 1 Week 12
Tmax for cabotegravir (Part 2 Injection 2) | Injection 2 Day 1 to Week 52 follow-up
Area under the concentration - time curve from time zero to last quantifiable time point (AUC[0-t]) for cabotegravir (Part 1 Injection 1) | Injection 1 Day 1 to Injection 1 Week 4
AUC(0-t) for cabotegravir (Part 1 Injection 2) | Injection 2 Day 1 to Injection 2 Week 4
AUC(0-t) for cabotegravir (Part 2 Injection 1) | Injection 1 Day 1 to Injection 1 Week 12
AUC(0-t) for cabotegravir (Part 2 Injection 2) | Injection 2 Day 1 to Injection 2 Week 12
Trough concentrations (Ctau) for cabotegravir (Part 1 Injection 1) | Injection 1 Day 1 to Injection 1 Week 4
Ctau for cabotegravir (Part 1 Injection 2) | Injection 2 Day 1 to Injection 2 Week 4
Ctau for cabotegravir (Part 2 Injection 1) | Injection 1 Day 1 to Injection 1 Week 12
Ctau for cabotegravir (Part 2 Injection 2) | Injection 2 Day 1 to Injection 2 Week 12
Apparent terminal phase half-life (T1/2) for cabotegravir (Part 1 Injection 2) | Injection 2 Week 4 to Week 52 follow-up
T1/2 for cabotegravir (Part 2 Injection 2) | Injection 2 Week 12 to Week 52 follow-up
Absorption rate constant (KALA) for cabotegravir (Part 1 Injection 2) | Injection 2 Week 4 to Week 52 follow-up
KALA for cabotegravir (Part 2 Injection 2) | Injection 2 Week 12 to Week 52 follow-up
Geometric mean ratio of plasma Ctau of CAB for Cohorts 1,2,3,4, 4b & 4h at Week4 (Part 1 Injection 1) compared to historical data of CAB 200 mg/mL IM (gluteus medius) (Week 8 Ctau following first injection at Week 4 in ATLAS [201585]/FLAIR [201584]Study) | At Injection 1 Week 4
Geometric mean ratio of plasma Ctau of CAB for Cohorts 1,2,3,4, 4b at Week 4 (Part 1 Injection 2) compared to historical data of CAB 200 mg/mL IM (gluteus medius) (Week 12 Ctau following first injection at Week 8 in ATLAS [201585]/FLAIR [201584]Study) | At Injection 2 Week 4
Geometric mean ratio of plasma Ctau of CAB for Cohorts 5 and 6 at Week 12(Part 2 Injection 1) compared to historical data of CAB 200 mg/mL IM (gluteus medius) (Week 8 Ctau following first injection at Week 4 in ATLAS [201585]/FLAIR [201584]Study) | At Injection 1 Week 12
Geometric mean ratio of plasma trough concentration (Ctau) of cabotegravir at Week 4 (Part 1 Injection 1) for each pairwise comparison between Cohorts 1, 2, 3, 4, 4b and 4h | At Injection 1 Week 4
Geometric mean ratio of plasma trough concentration (Ctau) of cabotegravir at Week 4 (Part 1 Injection 2) for each pairwise comparison between Cohorts 1, 2, 3, 4 and 4b | At Injection 2 Week 4
Geometric mean ratio of Plasma AUC(0-t) of cabotegravir at Week 4 (Part 1 Injection 1) for each pairwise comparison between Cohorts 1, 2, 3, 4, 4b and 4h | At Injection 1 Week 4
Geometric mean ratio of Plasma Cmax of cabotegravir at Week 4 (Part 1 Injection 2) for each pairwise comparison between Cohorts 1, 2, 3, 4 and 4b | At Injection 2 Week 4
Geometric mean ratio of Plasma Cmax of cabotegravir at Week 4 (Part 1 Injection 1) for each pairwise comparison between Cohorts 1, 2, 3, 4, 4b and 4h | At Injection 1 Week 4
Geometric mean ratio of Plasma AUC(0-t) of cabotegravir at Week 4 (Part 1 Injection 2) for each pairwise comparison between Cohorts 1, 2, 3, 4 and 4b | At Injection 2 Week 4

SECONDARY OUTCOMES:
Parts 1 and 2: Number of participants with adverse events (AEs) | Up to 52 weeks follow-up
Number of participants with liver biochemistry abnormalities | Up to 52 weeks follow-up
Cmax for cabotegravir following oral 30 mg administration | Up to Day 29
Tmax for cabotegravir following oral 30 mg administration | Up to Day 29
AUC(0-t) for cabotegravir following oral 30 mg administration | Up to Day 29
Concentration at 24 hours (C24) for cabotegravir following oral 30 mg administration | At 24 hours
Ctau for cabotegravir at Day 29 following oral 30 mg administration | Up to Day 29
Cmax of cabotegravir for cohort 4h | Injection 1 Day 1 to Week 52 follow-up
Tmax of cabotegravir for cohort 4h | Injection 1 Day 1 to Week 52 follow-up
AUC(0-t) of cabotegravir for cohort 4h | Injection 1 Day 1 to Week 52 follow-up
Ctau of cabotegravir for cohort 4h | Injection 1 Day 1 to Week 52 follow-up
T1/2 of cabotegravir for cohort 4h | Injection 1 Day 1 to Week 52 follow-up
KALA of cabotegravir for cohort 4h | Injection 1 Day 1 to Week 52 follow-up

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (5):
- United States (4):
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Berlin, New Jersey
  - GSK Investigational Site, Austin, Texas
- GSK Investigational Site, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com